CLINICAL TRIAL: NCT07374952
Title: Minimum Effective Volume of Lidocaine for Double-Injection Ultrasound-Guided Costoclavicular Block
Brief Title: Minimal Effective Volume 90% for Double-injection Costoclavicular Block
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Julián Aliste, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: COSTOCLAV DF 2026-11651
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Brachial Plexus Block, Lidocaine, Nerve Block
Keywords: Brachial plexus block, Lidocaine, nerve block

STUDY DESIGN:
Intervention Model Description: Dose finding study with an up-and-down methodology
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A research assistant (a licensed anesthesiologist) will prepare the local anesthetic solutions according to the sequential allocation. The operator, patient, and outcome assessor will remain blinded to the assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costoclavicular block with same previous successful volume (Active Comparator): Patients randomized to this group will receive the same volume that was successful in the previous recruitment.
  Interventions: Procedure: Ultrasound-guided double-injection costoclavicular nerve block with same previous volume
- Costoclavicular block with lower volume (Experimental): This group will be randomized to receive a fixed lower volume than the previously successful block.
  Interventions: Procedure: Ultrasound-guided double-injection costoclavicular nerve block with lower volume

INTERVENTIONS:
Procedure: Ultrasound-guided double-injection costoclavicular nerve block with same previous volume — ultrasound-guided double-injection costoclavicular nerve block with the same volume used in the previous successful block
  Arms: Costoclavicular block with same previous successful volume
Procedure: Ultrasound-guided double-injection costoclavicular nerve block with lower volume — Ultrasound-guided double-injection costoclavicular nerve block with lower volume than the previous successful block
  Arms: Costoclavicular block with lower volume

SUMMARY:
In 2020, a trial demonstrated that a 2-injection technique constitutes the optimal method for the costoclavicular block.

This study aims to determine the minimum amount of medication required to achieve a successful double-injection costoclavicular nerve.

Block dose assignment will be done using an up-and-down sequential method, called the Biased Coin Design (BCD).

The double-injection technique for US-guided costoclavicular block consists in depositing two thirds of the LA volume in the deep compartment (to anesthetize the posterior and medial cords), and one third of the injectate in the superficial compartment (to anesthetize the lateral cord).

The ED90 will be calculated using isotonic regression with a 95% confidence interval derived by bootstrapping.

DETAILED DESCRIPTION:
With the approval of the ethics committee of McGill University Health Centre, a total of 60 patients undergoing upper extremity surgery (elbow or below elbow) will be recruited.

The costoclavicular block will be performed under direct US vision until the tip is between the medial cord and the axillary artery. Two thirds of the volume of LA will be injected in this first location. Subsequently, the needle will be advanced until its tip is positioned next to the lateral cord. The remaining third of the LA volume will be injected in this second location.

Dose assignation will be done using an up-and-down sequential method, where the dose of each subsequent patient depends on the response of the previous patient, called the Biased Coin Design. The first subject recruited will receive a total of 30 mL of lidocaine 1.5 % with epinephrine 1: 200 000. Injection will be carried out by slow increments (5 mL) with negative aspiration between each increment.

The assignment of each subsequent dose will be based on the response of the previous patient as follows: if the previous patient did not have a successful block, the patient will receive the next higher dose, which is the previous dose incremented by 3.0 ml (i.e., an increment of 2.0 mL between the medial cord and the axillary artery, and an increment of 1.0 mL next to the lateral cord). If the previous patient had a successful block, the patient will be randomized to either receive the next lower dose, which is the previous dose decremented by 3.0 ml (i.e., a decrement of 2.0 mL between the medial cord and the axillary artery, and a decrement of 1.0 mL next to the lateral cord), with a probability b = 0.11, or to receive the same previous dose, with a probability 1 - b = 0.89. These are the probabilities required for assigning doses under the BCD for estimating ED90. A maximal dose of 40 mL will not be exceeded to avoid LA toxicity. If the previous patient did not respond and had been given the maximal dose the patient will also get the maximal dose. As soon as we recruit 45 patients with random dose assignment, we will terminate the enrollment procedure.

A research assistant will prepare and administer the injectate using syringes connected to the block needle. The operator and the patient will be blinded to the volume injected.

After LA injection at the second site, a catheter will be advanced 3 cm past the needle tip and secured to the skin. The purpose of the catheter is to allow LA supplementation for unsuccessful blocks, LA reinjection for lengthy surgical procedures or postoperative LA infusion for pain control.

The primary outcome is success rate which is defined as a minimal composite score of at least 14 points (out of a maximum of 16) is achieved at 30 minutes. The ED90 will be calculated using isotonic regression with a 95% confidence interval derived by bootstrapping .

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 30

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets≤ 100, International Normalized Ratio≥ 1.4 or partial prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases≥ 100)
* Allergy to LA
* Pregnancy
* Prior surgery in the infraclavicular region
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate | 30 minutes
  The primary outcome is success rate evaluated by the sensorimotor block which is defined as a minimal composite score of at least 14 points (out of a maximum of 16) is achieved at 30 minutes.
  The sensorimotor block will be assessed every 5 minutes until 30 minutes after the end of local anesthetic injection using a 16-point composite score evaluating sensory and motor block of musculocutaneous, median, radial, and ulnar nerves.
  Sensation will be assessed with ice in each nerve territory with a 0 to 2 point scale. 0= no block, patients can feel cold; 1= analgesic block, the patient can feel touch but not cold; 2= anesthetic block, the patient cannot feel cold or touch.
  The motor function will be assessed for each nerve with a 0 to 2 points scale where 0= no motor block; 1= paresis; 2= paralysis.
  Successful blocks at 30 minutes correlate with a final score ( sum of all individual sensory and motor scores) of at least 14 points out of 16.

SECONDARY OUTCOMES:
Operator level of experience | 1 hour before surgery
  expert vs. trainee
The number of needle passes | 1 hour before surgery
  The number of times the needle had to be withdrawn by ≥1 cm before redirecting to achieve the final position for local anesthetic injection.
Block performance time | 1 hour before surgery
  Sum of: 1- the acquisition time of the ultrasonographic image. and 2- the time to perform the block itself (from the skin anesthesia to the end of local anesthetic injection)
Block onset time | 1 hour before surgery
  Time required to reach a minimal sensorimotor composite score of 14 points out of a maximum of 16 points. The sensorimotor score is described in primary outcome.
Total anesthesia-related time | 1 hour before surgery
  Sum of: 1- the performance time and 2- the onset time
Intensity of pain during block procedure | 1 hour before surgery
  Evaluated with the Numeric Rating Scale for Pain. This scale is graduated from 0 to 10 points. A 0-point score represents the absence of pain, and a 10-points score represents the worst imaginable pain. Patients will be asked to rate their pain verbally with this scale. The blinded assessor will register the score reported.
Phrenic nerve block | 1 hour after arrival to post anesthesia care unit
  presence of dyspnea in postanesthetic care unit

OTHER OUTCOMES:
Incidence of nerve block side effects | From skin anesthesia to 60 minutes after the nerve block
  The presence of Horner syndrome, paresthesia, vascular puncture, hematoma, pneumothorax, or local anesthetic systemic toxicity after the nerve block.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stylianou M, Flournoy N. Dose finding using the biased coin up-and-down design and isotonic regression. Biometrics. 2002 Mar;58(1):171-7. doi: 10.1111/j.0006-341x.2002.00171.x. PMID 11890313
- [Background] Durham SD, Flournoy N, Rosenberger WF. A random walk rule for phase I clinical trials. Biometrics. 1997 Jun;53(2):745-60. PMID 9192462
- [Background] Saranteas T, Finlayson RJ, Tran DQH. Dose finding methodology for peripheral nerve blocks. Reg Anesth Pain Med. 2014;39:550-5.
- [Background] Layera S, Aliste J, Bravo D, Fernández D, Garcia A, Finlayson RJ, Tran DQ. Single- versus double-injection costoclavicular block: A randomized comparison. Reg Anesth Pain Med. 2020;45:209-13.
- [Background] Li JW, Songthamwat B, Samy W, Sala-Blanch X, Karmakar MK. Ultrasound-Guided Costoclavicular Brachial Plexus Block: Sonoanatomy, Technique, and Block Dynamics. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):233-240. doi: 10.1097/AAP.0000000000000566. PMID 28157792
- [Background] Karmakar MK, Sala-Blanch X, Songthamwat B, Tsui BC. Benefits of the costoclavicular space for ultrasound-guided infraclavicular brachial plexus block: description of a costoclavicular approach. Reg Anesth Pain Med. 2015 May-Jun;40(3):287-8. doi: 10.1097/AAP.0000000000000232. No abstract available. PMID 25899958